CLINICAL TRIAL: NCT00149435
Title: Cardiovascular Health Study (CHS) Events Follow-up Study
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Bruce Psaty, Professor, Medicine and Epidemiology, University of Washington
Other Study IDs: 1295; 5R01HL080295-07 (NIH)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Cerebrovascular Accident; Diabetes Mellitus; Heart Diseases; Hypertension; Heart Failure, Congestive
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Stroke; Diabetes Mellitus; Heart Diseases; Hypertension; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To support follow-up for the Cardiovascular Health Study (CHS) of coronary heart disease and stroke risk factors in adults 65 years or older.

DETAILED DESCRIPTION:
BACKGROUND:

The Cardiovascular Health Study (CHS) is an NHLBI-funded cohort study of risk factors for coronary heart disease (CHD) and stroke in adults 65 years or older. In the early 1990s, 5888 participants underwent examinations that included traditional risk factors and measures of sub-clinical disease. During follow-up, many exam components were repeated, and CVD events were ascertained. The National Heart, Lung, and Blood Institute has extended CHS contract funding (1) to implement a model for a transition from contract-funding to investigator-initiated research and (2) to enhance access to CHS data for future papers and ancillary studies by CHS and non-CHS colleagues. The Events Follow-up Study will provide a foundation for the transition. Current and future papers and ancillary studies using CHS data or stored specimens will have additional power and can be conducted more efficiently if a service events-core continues to collect and adjudicate CVD events and deaths in a standardized fashion.

DESIGN NARRATIVE:

Structurally, the primary aims are: (1) to evaluate the incidence rates of and risk factors for CVD in older adults, including comparisons between blacks and whites, men and women, young old and old; (2) the evaluation of prognosis in inception cohorts of older adults with new-onset conditions such as heart failure (HF) and atrial fibrillation; and (3) the evaluation of associations between risk-factor change and the incidence of subsequent events. Questions of interest include: What are the determinants of the low CHD incidence in women 80 yrs and older? Do older black women also have a low CHD incidence? What are the determinants of CHD, HF, and stroke in adults 80 and older? Are risk factors different between men and women, whites and blacks? Do traditional risk factors and measures of sub-clinical disease continue to be powerful predictors of CHD, HF and stroke in those 80 and older? In this study, the investigators expect to make over 20,000 phone calls to identify 6000 hospitalizations, 1000 deaths, 3000 events for detailed review, and 1500 new events, including 370 CHD, 300 stroke, and 450 HF. These new events represent an increase in the number of CVD events of 29% to 35% in whites and an increase of 40% to 49% in blacks. The data and specimens collected in CHS represent a major national resource for the study of health, aging, and cardiovascular disease in older adults. Additional events follow-up will not only provide the opportunity to address the aims of this study, but also enhance the power of current and future CHS papers and ancillary studies by CHS and non-CHS colleagues.

ELIGIBILITY:
No eligibility criteria

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 5888 (Actual)
Dates: Start 2005-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Cardiac health | Annual
  Incidence of cardiac related death

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Psaty, Study Director — University of Washington

REFERENCES:
- [Derived] Fretts AM, Follis JL, Nettleton JA, Lemaitre RN, Ngwa JS, Wojczynski MK, Kalafati IP, Varga TV, Frazier-Wood AC, Houston DK, Lahti J, Ericson U, van den Hooven EH, Mikkila V, Kiefte-de Jong JC, Mozaffarian D, Rice K, Renstrom F, North KE, McKeown NM, Feitosa MF, Kanoni S, Smith CE, Garcia ME, Tiainen AM, Sonestedt E, Manichaikul A, van Rooij FJ, Dimitriou M, Raitakari O, Pankow JS, Djousse L, Province MA, Hu FB, Lai CQ, Keller MF, Perala MM, Rotter JI, Hofman A, Graff M, Kahonen M, Mukamal K, Johansson I, Ordovas JM, Liu Y, Mannisto S, Uitterlinden AG, Deloukas P, Seppala I, Psaty BM, Cupples LA, Borecki IB, Franks PW, Arnett DK, Nalls MA, Eriksson JG, Orho-Melander M, Franco OH, Lehtimaki T, Dedoussis GV, Meigs JB, Siscovick DS. Consumption of meat is associated with higher fasting glucose and insulin concentrations regardless of glucose and insulin genetic risk scores: a meta-analysis of 50,345 Caucasians. Am J Clin Nutr. 2015 Nov;102(5):1266-78. doi: 10.3945/ajcn.114.101238. Epub 2015 Sep 9. PMID 26354543